CLINICAL TRIAL: NCT03901794
Title: Relationship Between Hemodynamic Change and Fluid Removed During Hemodialysis Measured by Non-invasive Monitor
Brief Title: Relationship Between Hemodynamic Change and Fluid Removed During Hemodialysis
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201702064RIPB
Record Dates: First submitted 2019-03-11; First posted 2019-04-03 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2017-04

CONDITIONS: Hemodialysis Complication; Hemodialysis-Induced Symptom

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- With Clear Sight: record and observe the data including SVI, CI, SVR with clearSight during hemodialysis
  Interventions: Device: Non-invasive hemodynamic monitor

INTERVENTIONS:
Device: Non-invasive hemodynamic monitor — MAP, HR, CO, SVI, from Non-invasive hemodynamic monitor

SUMMARY:
Relationship between hemodynamic change and fluid removed during hemodialysis measured by non-invasive monitor

DETAILED DESCRIPTION:
By applying non-invasive hemodynamic monitors (ex. ClearSight, I-COM), the trends of mean arterial pressure (MAP), stroke volume (SV), cardiac index (CI) and calculated systemic vascular resistance (SVR) were collected along with volume removal by hemodialysis on ESRD patients. All data were compared and analyzed to detect the sequential body volume status as well as the autonomic responses during hemodialysis.

ELIGIBILITY:
Inclusion criteria:

1. Patients who were schedured with regular hemodialysis for end-stage renal disease.

Exclusion criteria:

1. Emergent hemodialysis
2. Medical conditions with poor peripheral circulation such as Raynaud's disease or PAOD
3. Skin defects or wounds over area to be applied for measurement (Wrist and fingers)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: end-stage renal disease patients who were under regular hemodialysis
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-05-06 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
fluid removed along with hemodialysis | 4 hours
  the fluid volume removed from hemodialysis (mL/hour),
changes of mean arterial pressure along with hemodialysis | 4 hours
  record of mean arterial pressure (mmHg) per 30 minutes
changes of heart rate along with hemodialysis | 4 hours
  record of heart rate (beats/ minute) per 30 minutes
changes of stroke volume along with hemodialysis | 4 hours
  record of stroke volume (SV, (mL/ beat)per 30 minutes
changes of cardiac output along with hemodialysis | 4 hours
  record of cardiac output ( liter/ minute)per 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: ST Chen, Study Chair — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lai CJ, Shih CC, Huang HH, Chien MH, Wu MS, Cheng YJ. Detecting Volemic, Cardiac, and Autonomic Responses From Hypervolemia to Normovolemia via Non-Invasive ClearSight Hemodynamic Monitoring During Hemodialysis: An Observational Investigation. Front Physiol. 2022 Apr 28;13:775631. doi: 10.3389/fphys.2022.775631. eCollection 2022. PMID 35574491